CLINICAL TRIAL: NCT06256419
Title: Department of Pharmacy, the Affiliated Hospital of Xuzhou Medical University
Brief Title: Association of Gene Polymorphism With Susceptibility to T2DM and the Therapeutic Responses to Exenatide in Chinese Patients With T2DM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Affiliated Hospital of Xuzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: XYFY2023-KL479-01
Record Dates: First submitted 2024-02-05; First posted 2024-02-13 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Type 2 Diabetes Mellitus; Susceptibility, Genetic
Keywords: Type 2 Diabetes Mellitus; GLP-1 RA; gene polymorphism; susceptibility gene; variation
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Genetic Predisposition to Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- efficacy difference of GLP-1RA (Experimental): Responders group and non-responders group
  Interventions: Drug: GLP-1 receptor agonist; Drug: responders group and nonresponders group

INTERVENTIONS:
Drug: GLP-1 receptor agonist — Eligible patients with T2DM were required to have received GLP-1RA as monotherapy or in combination with other antidiabetic agents. GLP-1 RA was injected subcutaneously at standard dose and frequency for consecutive 6 months in patients with T2DM.
Drug: responders group and nonresponders group — For all the patients with type 2 diabetes who were initially enrolled in the study, blood samples were obtained for genotyping before the administration of GLP-1 receptor agonists. Patients were re-screened according to whether they had used GLP-1 RA continuously for more than 6 months and had completed the specified follow-up tasks.
  Patients were divided according to the type of T2DM susceptibility genes. Or all were divided into responses group and nonresponses group according to whether they had glycemic response (△HbA1c↓ ≥1.0%) and weight response (△weight↓ ≥3.0%) after taking GLP-1 receptor agonist for 6 months.
  According to the above grouping, the variables that can predict the efficacy of the drug were identified, and the weight of the influence of these variables on the efficacy was evaluated.

SUMMARY:
This is a retrospective cohort study of patients with T2DM who were treated with exenatide twice daily as a part of their diabetes care for at least 12 months. The objective of this study is to investigate the influence of T2DM susceptibility gene polymorphisms (NOS1AP, KCNQ1, TCF7L2, WSF1, GLP-1R, etc.) on the efficacy of GLP-1 RA (exenatide, liraglutide, etc.), to identify the variables that can predict the efficacy of GLP-1 RA, and to evaluate the weight of these variables on the efficacy.

DETAILED DESCRIPTION:
T2DM is a polygenic genetic disease. The individual differences in the efficacy of antidiabetic drugs are caused by the cumulative effect of multiple gene polymorphisms, and are related to environmental factors and lifestyle. The results of single gene polymorphism cannot fully explain the individual differences in the efficacy of antidiabetic drugs. Verifying the correlation between T2DM gene polymorphisms and the efficacy of antidiabetic drugs, clarifying the genetic determinants of individual differences in the efficacy of antidiabetic drugs, and predicting the efficacy and side effects of antidiabetic drugs are of great significance for the formulation of precise medication regimens for T2DM patients.

Many guidelines recommend the preferential use of GLP-1 RA after single drug or multiple oral hypoglycemic drugs and basic insulin therapy for poor glycemic control. However, the clinical responsiveness to GLP-1 RA varies among patients with T2DM. It has been reported that genetic factors are the important reasons for individual variation in therapeutic response of antidiabetic drugs. At present, dozens of gene loci related to therapeutic response of antidiabetic drugs have been screened, which are of great clinical significance in guiding clinical individualized treatment, improving the efficacy and safety of drugs, and reducing the drug costs.

GLP-1 RA was injected subcutaneously at standard dose and frequency for consecutive 6 months. The patients were visited at moths 0, 3, and 6, and medical histories, physical examinations, and routine clinical laboratory tests were performed during these visits. The general anthropometric parameters considered for this study were height (m), weight (kg), and waist and hip circumferences (cm) at baseline, 3 months and 6months after exenatide treatment.

Patients who had an HbA1c reduction ≥1.0% or HbA1c <7.0% after exenatide treatment for six consecutive months were considered responders, while patients who failed to achieve this decrease were considered non-responders. The clinical data were collected and analyzed to determine the variables that could predict the efficacy of GLP-1 RA, and to evaluate the weight of the influence of these variables on the efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. a diagnosis of T2DM
2. a body mass index (BMI) of 20-35 kg/m2
3. an HbA1c of 7.0%-12%, an age of 25-70 years
4. required data available at baseline and 6 months after GLP-1RA therapy.

Exclusion Criteria:

1. Patients with serious diseases such as acute myocardial infarction, cerebral vascular accident, trauma, kidney or liver diseases, severe gastrointestinal dysfunction, and history of pancreatitis
2. patients receiving GLP-1 analogues, weight loss drugs, glucocorticoids, drugs affecting gastrointestinal peristalsis in the past 3 months
3. those with missing data at the time points of baseline, 3 months, and 6 months after GLP-1 RA therapy.

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2028-01-31 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline HbA1c and baseline weight at 6 month | 6 month after GLP-1 RA treatment
  In order to observe the change from baseline HbA1c and baseline weight at 6 month after GLP-1 RA treatment
To identify and evaluate the variable factors influencing GLP-1 RA efficacy | 1 month after sample integration
  The variable factors that predict the efficacy of GLP-1 RA were identified and the weight these variables on the efficacy was assessed
Genotype identification in patients with T2DM | 1 month after sample collecting
  Blood samples were collected from T2DM patients for genotyping

SECONDARY OUTCOMES:
Incidence and severity of possible adverse reaction within 6 month after GLP-1 RA treatment | 6 months after GLP-1 RA treatment
  To evaluate the incidence and severity of possible adverse reaction within 6 month after GLP-1 RA treatment, including gastrointestinal reaction and hypoglycemia

CONTACTS AND LOCATIONS:
Locations (1):
- China, Jiangsu, Department of Endocrinology, Xuzhou, China, China

IPD SHARING:
Plan to Share IPD: No